CLINICAL TRIAL: NCT06087549
Title: PENG Block vs. ESP Block for Pediatric Hip Surgery. A Randomized, Prospective Double-blinded Clinical Trial.
Brief Title: PENG Block vs. ESP Block for Pediatric Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4/2023
Record Dates: First submitted 2023-07-05; First posted 2023-10-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hip Dysplasia; Hip Injuries; Hip Fractures; Hip Disease
MeSH Terms: conditions — Hip Dislocation; Hip Injuries; Hip Fractures | interventions — Ropivacaine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Three groups:
  Group I -control Group II - PENG block Group III - ESP block
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly allocated to receive ultrasound-guided PENG block, ESP block, or only spinal anesthesia by computer software 1:1:1. A researcher who will not involve in the study will prepare the randomization list and concealed group assignments in consecutively numbered, sealed, opaque envelopes. A consultant anesthesiologist will follow management to open the envelopes shortly before the nerve block performance to reveal the group allocation and perform the procedure according to the assignment. The patients and their anesthesia team, surgeon, operating room staff, and parents will be masked to the study group allocation. Group blinding unmasking will only occur once the statistical analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): regional anesthesia: spinal anesthesia - 0,1ml/kg 0,5% ropivacaine
  Interventions: Other: Standard care
- Pericapsular nerve group block (PENG) group (Active Comparator): regional anesthesia: spinal anesthesia - 0,1ml/kg 0,5% ropivacaine + PENG block - 0.5mL/kg 0.2% ropivacaine, max. 20mL
  Interventions: Drug: Pericapsular nerve group block using 0.2% ropivacaine
- Erector Spinae Plane Block (ESPB) group (Active Comparator): regional anesthesia: spinal anesthesia - 0,1ml/kg 0,5% ropivacaine + ESP block - 0.5mL/kg 0.2% ropivacaine, max. 20mL
  Interventions: Drug: Erector Spinae Plane Block using 0.2% ropivacaine

INTERVENTIONS:
Drug: Pericapsular nerve group block using 0.2% ropivacaine — Unilateral ultrasound guided pericapsular nerve block using 0.5mL/kg 0.2% Ropimol (max 20mL)
  Arms: Pericapsular nerve group block (PENG) group
Drug: Erector Spinae Plane Block using 0.2% ropivacaine — Unilateral ultrasound guided erector spinae block using 0.5mL/kg 0.2% Ropimol (max 20mL)
  Arms: Erector Spinae Plane Block (ESPB) group
Other: Standard care — No erector spinae block and no pericapsular nerve group block
  Other Names: No erector spinae block and no pericapsular nerve group block
  Arms: Control group

SUMMARY:
The study compares the effectiveness and safety of the pericapsular nerve blockade vs. ESPB in pediatric patients who underwent hip surgeries.

DETAILED DESCRIPTION:
The study compares the effectiveness and safety of the pericapsular nerve blockade vs. ESPB in pediatric patients who underwent hip surgeries. In addition, we aim to determine the optimal volume of local anesthetics needed to achieve a satisfactory level of analgesia.

ELIGIBILITY:
Inclusion Criteria:

- pediatric patients aged between 0-12 years who will undergo hip surgery

Exclusion Criteria:

* a history of chronic pain use of gabapentin/pregabalin for > 3 months opioid use > 1 repeated opioid prescription in the last three months
* morbid obesity (BMI > 99th percentile)
* Infection at block application area
* coagulopathy

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
FLACC score | 48 hours after surgery
  The FLACC scale or Face, Legs, Activity, Cry, Controllability Scale is used to assess pain for children between the ages of 2 months and seven years or individuals unable to communicate their pain. The scale is scored in a range of 0-10, with 0 representing no pain.

SECONDARY OUTCOMES:
NLR | 48 hours after surgery
  neutrophil-to-lymphocyte ratio
PLR | 48 hours after surgery
  platelet-to-lymphocyte ratio
total opioid consumption | 48 hours after surgery
  morphine equivalents in miligrams

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, Prof.dr hab, Study Chair — Poznań University of Medical Sciences
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland